CLINICAL TRIAL: NCT01483846
Title: A Phase 1b, Single-Site, Randomized, Double-Blind,Placebo-Controlled, Dose-Escalation Study: Safety, Pharmacokinetics, and Antihyperalgesic Activity of Multiple Doses of AV-101 on Capsaicin-Induced Pain in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Doses of AV-101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VistaGen Therapeutics, Inc. (Industry)
Collaborators: Cato Research (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VSG-CL-002; R44DA018515 (NIH)
Record Dates: First submitted 2011-11-16; First posted 2011-12-01 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic Pain; Capsaicin Induced Pain
MeSH Terms: conditions — Neuralgia | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AV-101 (Experimental): Subjects will be randomized into one of three dose cohorts (360, 1,080, and 1,440 mg) to receive a daily oral dose for 14 consecutive days. Each cohort will have 12 subjects on active drug and 4 subjects on placebo.
  --------------------------------------------------------------------------------
  Interventions: Drug: AV-101
- microcrystalline cellulose (Placebo Comparator): Subjects will be randomized into one of three cohorts (360, 1,080, and 1,440 mg) to receive a daily oral dose for 14 consecutive days. Each cohort will have 12 subjects on active drug and 4 subjects on placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AV-101 — Placebo or AV-101 at 360 mg, 1080 mg, or 1440 mg will be dosed once daily for 14 consecutive days.
  Other Names: L-4-Cl-KYN
  Arms: AV-101
Drug: Placebo — Placebo or AV-101 at 360 mg, 1080 mg, or 1440 mg will be dosed once daily for 14 consecutive days.
  Other Names: microcrystalline cellulose
  Arms: microcrystalline cellulose

SUMMARY:
This is a Phase 1b study involving multiple oral doses of AV-101 in healthy male and female subjects. The safety, pharmacokinetics, and antihyperalgesic effect of AV-101 on capsaicin-induced hyperalgesia will be assessed.

DETAILED DESCRIPTION:
Healthy subjects will be randomized into three dose cohorts (360, 1,080, and 1,440 mg) to receive daily oral doses of AV-101 for 14 consecutive days. Each cohort has 12 subjects on active drug and 4 subjects on placebo. Safety, PK, and antihyperalgesic effects of treatment with AV-101 will be assessed.

At the screening visit between Day -28 and Day -7 before randomization, 250 μg of capsaicin will be intradermally delivered into the volar aspect of one forearm. Subjects must report a pain score of at least 4 out of 10 to qualify for the study. On Day 1 and Day 14 the following data are collected: (1) neurosensory testing (thermal sensation, thermal pain, touch, and mechanical pain) on the forearm; (2) neurocognitive evaluation; and (3) 12-lead electrocardiogram, blood pressure, heart rate, respiratory rate, and temperature. PK samples will be collected on Days 1, 2, 14, and 15. The capsaicin-induced pain will be assessed at screening, on Day 1, and Day 14. An intradermal injection of capsaicin into the forearm on Day 1 and Day 14 will be followed by the efficacy measures. On Day 1 before administration of the first dose, subjects will be given a paper diary to record daily self-administration of each dose, concomitant medications, and adverse events during the 14-day treatment period.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for participation in the full study only if all of the following criteria are met:

  1. Be male or female, aged 21 to 60 years inclusive, healthy, able and willing to provide written informed consent to participate in the study.
  2. Be able to read and speak English sufficiently to understand and follow the study instructions, including completion of pain intensity rating scales.
  3. For males, must use birth control (condom) to prevent fathering children; for females must be nonlactating, not pregnant, and using a reliable contraception method (e.g., abstinence, intrauterine device, hormonal birth control, or double barrier method [male condom, female condom, or diaphragm plus a spermicidal agent such as contraceptive foam, jelly, or cream]).
  4. Have a visual analog pain score of at least 4 out of 10 at screening.

Exclusion Criteria:

* Subjects will be excluded from the study if any one or more of the following conditions apply:

  1. History of peripheral neuropathy or any chronic pain condition.
  2. History of significant hepatic, ophthalmic (including previous or current cataract), cardiovascular, renal, gastrointestinal, hematological, neurological, endocrine (including diabetes), metabolic, pulmonary, or psychiatric disease. Significance will be determined by the principal investigator.
  3. Clinically significant abnormality on the screening electrocardiogram that in the judgment of the investigator would place the subject at risk of cardiac adverse event as a result of capsaicin injection or administration of AV-101.
  4. Cognitive or psychiatric disorders that may diminish compliance with study procedures.
  5. Dermatopathology, skin hypersensitivity, or skin lesions in the areas of capsaicin application.
  6. Allergy to capsaicin or the study medication.
  7. Current tobacco use.
  8. Use of chemotherapy agents or history of cancer, other than resolved skin cancer, within 5 years before the screening visit.
  9. History of drug or alcohol abuse within 1 year before screening.
  10. History of AIDS, testing as HIV positive, or use of antiretroviral therapy.
  11. Use of, within 4 weeks before study drug dosing, any investigational drug, any epidural or intrathecal agent, corticosteroids, topical anesthetics, topical analgesics, central alpha agents (e.g., clonidine), alpha blockers (e.g., praxosin, terazosin), beta blockers, calcium channel blockers, or ACE inhibitors.
  12. Use within 7 days before and during the entire period of study drug dosing of long-acting nonsteroidal anti-inflammatory drug (NSAIDs) such as piroxicam or naproxen.
  13. Use within 36 hours before and during the entire period of study drug dosing of NSAIDs, aspirin, acetaminophen, antihistamines, sympathomimetics (e.g., pseudoephedrine and ephedrine), caffeine or alcohol.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | PK samples will be collected at time 0, 0.5, 1.5, 2, 4, 6, 8, 12, and 24 hours post-dosing on Day 1 and Day 14.
  To evaluate pharmacokinetics of three dose levels of orally-administered AV-101 given once a day for 14 days in healthy volunteers by measuring Cmax, half-life, Tmax, and AUC.
Safety | 28 days
  To evaluate the safety of three dose levels of orally-administered AV-101 given once a day for 14 days in healthy volunteers by evaluating the number of subjects with treatment-emergent adverse events and changes from baseline to end of study in vital signs, hematology, hepatic profile, renal profile, urinalysis, and clinical laboratory parameters.

SECONDARY OUTCOMES:
Antihyperalgesic activity | 28-49 Days
  To examine the antihyperalgesic effects of orally-administered, multiple doses of AV-101 in healthy volunteers by using the intradermal capsaicin model.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Snodgrass, PhD, Study Director — VistaGen Therapeutics, Inc.
Locations (1):
- UCSD Medical Center, San Diego, California, United States

REFERENCES:
- [Derived] Wallace M, White A, Grako KA, Lane R, Cato AJ, Snodgrass HR. Randomized, double-blind, placebo-controlled, dose-escalation study: Investigation of the safety, pharmacokinetics, and antihyperalgesic activity of l-4-chlorokynurenine in healthy volunteers. Scand J Pain. 2017 Oct;17:243-251. doi: 10.1016/j.sjpain.2017.05.004. Epub 2017 Jun 15. PMID 29229209